CLINICAL TRIAL: NCT04524559
Title: Feasibility Of Oral Sensorimotor Stimulation And Sequenced Trunk Co-Activation On Oropharyngeal Dysphagia In Children With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Feasibility Of Oral Sensorimotor Stimulation On Oropharyngeal Dysphagia In Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira M Abd-elmonem, PHD, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oral Sensorimotor Stimulation
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Physical Therapy
Keywords: Spastic Quadriplegia; Cerebral Palsy; Oropharyngeal Dysphagia; Oral Sensorimotor Stimulation
MeSH Terms: conditions — Quadriplegia; Cerebral Palsy; Deglutition Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy training (Placebo Comparator): received 90 minutes conventional physical therapy training focused on regaining typical movement, prohibiting abnormal muscle tone, promoting postural reactions and enhancing postural mechanisms.
  Interventions: Other: conventional physical therapy training
- oral stimulation (Experimental): received 30 minutes of oral motor training five days week. The training included oral stimulation (facilitation) conducted before the child's actual meal time. The designed protocol comprised modified perioral and intraoral maneuvers based on Fucile's protocol
  Interventions: Other: conventional physical therapy training; Other: oral motor training.

INTERVENTIONS:
Other: conventional physical therapy training — The program focused on regaining typical movement, prohibiting abnormal muscle tone, promoting postural reactions and enhancing postural mechanisms. The program was applied via certified physical therapists five days/week for 4 successive months. The intended goals of the treatment program were achieved through:
  * Neurodevelopmental based training (NDT)
  * Functional stretching exercises to preserve muscle and soft tissues elasticity
  * Sequenced trunk co-activation (STA) exercises
  * Righting and protective reactions It is worth mentioned that the exercises applied in each session was influenced by the age and the specific functional abilities within the selected activity.
  Other Names: Neurodevelopmental based training (NDT); Functional stretching exercises; Sequenced trunk co-activation (STA) exercises; - Righting and protective reactions:
Other: oral motor training. — Children in the experimental group received 30 minutes of oral motor training five days week. The training included oral stimulation (facilitation) conducted before the child's actual meal time.
  The designed protocol comprised modified perioral and intraoral maneuvers based on Fucile's protocol. The utmost aims of the protocol were to decrease hypersensitivity of oral structures, increase jaws movement, and reinforce muscle strength, improve tongue movement and enhance oral motor organization
  Arms: oral stimulation

SUMMARY:
Children with CP encounter swallow and feeding impairments, especially in infancy and childhood with long meal times with late development of oral motor skills resulting in poor growth.

DETAILED DESCRIPTION:
this study will be conducted to explore the feasibility of oral sensorimotor stimulation combined with sequenced trunk co-activation on oropharyngeal dysphagia in children with spastic quadriplegic CP.

ELIGIBILITY:
Inclusion criteria

* Diagnosed as spastic quadrilepgic CP
* Both genders
* Aged from 12 to 48 months
* Scored ≤ 10 on an initial evaluation of Oral Motor Assessment Scale.
* Having at least a problem of oral motor functions (drooling, swallowing, and/or sucking); independent feeding
* Grade ≥ 2 spasticity according to the MAS
* Level IV and V motor function according to the GMFCS-R&E.
* Partial head and trunk control. Exclusion criteria
* Gum and/or dental problems
* Congenital problems of mouth and soft plate
* Uncontrolled seizures
* Any metabolic disorders
* Cardiopulmonary disorders
* Significant mental problems.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Oral motor skills | period of the treatment was 4 successive months
  The Oral Motor Assessment Scale is a reliable and accurate scale frequently used to assess oral-motor skills in young patients with neurological disorders. It is a useful tool that can be used in assessment and interventional studies. The full assessment takes approximately 20 minutes to be completed for each child giving score as passive (0), sub-functional (1), semi-functional (2) and functional (3) with higher scores represent better oral-motor skills

SECONDARY OUTCOMES:
- Physical growth | period of the treatment was 4 successive months
  The body mass was measured via weight scale to detect the physical growth changes overtime.
- Segmental trunk control | period of the treatment was 4 successive months
  The Segmental Assessment of Trunk Control (SATCo) was applied to assess upright trunk postural control in sitting position. It is an ordinal scale with a grade 1 to 7 is assigned for each segment with the score 7 indicates that the infant can't retain independent sitting (no hand support). A score of 8 is given as full trunk control is gained. Each infant would therefore have three scores to represent the static, active and reactive trunk control (higher scores represent better trunk control)
- Gross motor function | period of the treatment was 4 successive months
  The motor function was conducted via the gross motor function measure (GMFM). The GMFM-88 is a valid and reliable observational criterion-referenced tool graded from 0-100 was developed to assess motor function in children with CP or Down syndrome. It measures gross motor function in five domains with 88 items with higher scores represent better motor function

CONTACTS AND LOCATIONS:
Overall Officials: sara s saad-Eldeen, Study Director — MTI university, Egypt
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No